CLINICAL TRIAL: NCT02914912
Title: Investigation of Chronic Intestinal Ischemia
Status: Active, not recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Syed Sajid Hussain Kazmi, Consultant Surgeon, Oslo University Hospital
Other Study IDs: 2016/682
Record Dates: First submitted 2016-09-14; First posted 2016-09-26 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Chronic Mesenteric Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- GALS symptomatic patients group: Patients with chronic mesenteric ischemia (CMI) symptoms shall be investigated with gastroscopy-assisted laser Doppler flowmetry and visible light spectroscopy.
  The examination will be performed before and after the surgical or endovascular treatment for CMI.
  Besides, the patients treated with either open or laparoscopic mesenteric bypass shall be examined during the operation with transserosal microcirculatory assessment of the stomach and duodenum using laser Doppler flowmetry and visible light spectroscopy.
- CMI caused by median arcuate ligament syndrome (MALS): Patients with chronic mesenteric ischemia (CMI) symptoms caused by MALS shall be investigated with gastroscopy-assisted laser Doppler flowmetry and visible light spectroscopy. The examination will be performed before and after the surgical or endovascular treatment for MALS.
  Besides, the patients treated with an either open or laparoscopic technique for MALS shall be examined during the operation with transserosal microcirculatory assessment of the stomach and duodenum using laser Doppler flowmetry and visible light spectroscopy.
- Healthy individuals without CMI or MALS: A group of healthy individuals with no symptoms of CMI or MALS shall be investigated with gastroscopy-assisted laser Doppler flowmetry and visible light spectroscopy.

SUMMARY:
Patients suspected of chronic mesenteric ischemia caused by atherosclerosis or median arcuate ligament syndrome shall be investigated with trans mucosal and transserosal laser Doppler flowmeter and visible light spectroscopy.

DETAILED DESCRIPTION:
Patients with suspected chronic mesenteric ischemia (included median arcuate ligament syndrome/truncus coeliacus compression syndrome) referred to the vascular surgery department for investigation of splanchnic and mesenteric circulation shall be included in this study.

In addition to CT angiography, patients shall be investigated

1. with gastroscopy-assisted laser Doppler flowmetry and light spectroscopy (GALS) before and after the surgical or endovascular treatment
2. Endoscopic ultrasound before and after the surgical or endovascular treatment
3. Transserosal laser Doppler flowmetry and light spectroscopy during the surgical treatment
4. Plasma Ischemia bio-markers, before and after the surgical or endovascular treatment
5. Health related quality of life assessed with EQ5D and SF36 before and after the treatment
6. clinical outcomes of the treatment (early and late results).

ELIGIBILITY:
Inclusion Criteria:

Clinical chronic mesenteric ischemia caused by either atherosclerosis or median arcuate ligament syndrome

Exclusion Criteria:

Patients unable to go through gastroscopy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients suspected of chronic mesenteric ischemia caused by either atherosclerosis or median arcuate ligament syndrome and confirmed with CTA, duplex ultrasound, and clinical examination shall be included in the study. The included patients are referred to the Department of Vascular Surgery for investigation and treatment of the CMI and MALS.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-09; Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Transmucosal Oxygen concentration of the stomach and duodenum | Baseline, 3 months and 12 months
  Repeated measurments at baseline 3, and 12 months after the surgical or endovascular treatment of chronic mesenteric ischemia (CMI) and median arcuate ligament syndrome (MALS) shall be performed. With the help of gastoscopy assisted Laser Doppler flowmeter and visible light spectroscopy, transmocosal SaO2, rHb concentration, flow and velocity in arbitrary units shall be measured.

SECONDARY OUTCOMES:
Ischemia biomarkers | 10 years
  Plasma levels of intestinal ischemia biomarkers, alpha glutathione s transeferase, intestinal fatty acid binding protein, human immune modified globulin and plasma citrolline shall be examined before and after the surgical or endovascular treatment of the patients with either open or laparoscopic surgery, or endovascular treatment. Blood samples from a cohort of healthy individuals without any symptoms of CMI or MALS shall be tested for the same ischemia biomarkers.
Health-related quality of life in the patients with chronic mesenteric ischemia | 10 years
  Quality of life assesment at baseline and after treatment with EQ-5D
Clinical outcomes of revascularization in the patients with chronic mesenteric ischemia | 10 years
  Chronic mesenteric ischemia and median arcuate ligament syndrome patients treated with either open/ laparoscopic vascular surgery or endovascular treatment shall be routinely followed-up at the out-patients department for the results of the treatment and the post operative complications, effect of revascularization on the mesenteric ischemia symptoms, patency of endovascular or open revascularization procedure. Routine clinical follow-up shall be 30 days post operatively, 3 months, 12 months and yearly thereafter. Besides the patency of the revascularized mesenteric artery will be determined with duplex ultrasound.
Transserosal microcirculation assessment | 10 years
  The patients with MALS and CMI treated with an either open or laparoscopic surgery shall be examined with transserosal Laser Doppler flowmetery and visible light spectroscopy of the stomach and duodenum during the operation. Transserosal SaO2, relative Hb concentration, blood flow and velocity in arbitrary units will be measured with the Laser doppler flowmeter and visible light spectroscope applaied directly to the surface of stomach and duodenum under the surgical procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Sajid Hussain Kazmi, MD PhD, Principal Investigator — Oslo University Hospital
Locations (2):
- Norway (2):
  - Oslo University Hospital, Oslo
  - Department of vascular surgery, Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: Yes
The PI can share anonymous study data after completion of the study.
Supporting Information: Study Protocol, ICF
Time Frame: Anonymous data can be available up to two years after completion of the study.
Access Criteria: Data will be shared with investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. Proposals should be directed to the principal investigator. To gain data access, data requesters will need to sign a data access agreement.